CLINICAL TRIAL: NCT02413996
Title: Effects of Virtual Reality Rehabilitation in Patients With Total Knee Arthroplasty: A Randomised Controlled Trial
Brief Title: Effects of Virtual Reality Rehabilitation in Patients With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Davide Tornese, Medico Chirurgo Specialista in Medicina Fisica e Riabilitazione, Specialista in Medicina dello Sport, Responsabile reparto di Riabilitazione Sportiva, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRRS
Record Dates: First submitted 2015-03-11; First posted 2015-04-10 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Total Knee Replacement; Virtual Reality Therapy; Osteoarthritis; Knee Arthroplasty; Rehabilitation
Keywords: Virtual Reality Therapy; Rehabilitation; Total Knee Replacement; Knee Arthroplasty; Exercise; Arthritis; Rheumatic Disease
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Arthritis; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: A phase III randomized clinical trial was approved by the San Raffaele Hospital's Ethic Committee of Milan (31/03/2014)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VRRS rehabilitation (Experimental): exercise therapy through a virtual reality rehabilitation system (VRRS) in addition to a knee continuous passive motion device ( Kinetec® continuous passive motion ( CPM )) and functional activities (e.g.,stairs, walking)
  Interventions: Device: Kinetec® knee continuous passive motion (CPM ); Behavioral: Functional activities; Other: VRRS rehabilitation
- traditional rehabilitation (Active Comparator): exercise therapy through a traditional rehabilitation training in addition to a knee continuous passive motion device ( Kinetec® continuous passive motion ( CPM )) and functional activities (e.g.,stairs, walking)
  Interventions: Device: Kinetec® knee continuous passive motion (CPM ); Behavioral: Functional activities; Other: traditional rehabilitation

INTERVENTIONS:
Device: Kinetec® knee continuous passive motion (CPM ) — CPM of the knee
Behavioral: Functional activities — Stairs, walking
Other: VRRS rehabilitation — exercise therapy through a virtual reality rehabilitation system (VRRS)
  Arms: VRRS rehabilitation
Other: traditional rehabilitation — exercise therapy through a traditional rehabilitation training made by physiotherapists
  Arms: traditional rehabilitation

SUMMARY:
The aim of this study is to assess the efficacy of virtual rehabilitation through the Virtual Reality Rehabilitation System (VRRS) versus traditional rehabilitation improving the functional outcomes after primary Total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
Following ethics approval by the Ospedale San Raffaele, 84 adults aged between 45 and 80 years old will be recruited for the study, excluding people with unstable serious disease (e.g., heart or lung disease), previous orthopedics pathologies on the same side (e.g., hip arthroprosthesis), pregnancy and intake of psychotropic drugs.

Patients who consent to participate in this study will be randomized into two rehabilitation groups after TKA: experimental (virtual rehabilitation) and control (traditional rehabilitation). In the experimental arm, subjects will undergo a virtual rehabilitation training during the post-surgical rehabilitation period, in addition to passive knee range of motion device (kinetec) and functional activity (stairs). In the control arm, subjects with similar demographic characteristics to those of the experimental arm, will undergo the usual physiotherapy rehabilitation, in addition to passive knee range of motion device (kinetec) and functional activity (stairs). Both control and study interventions will be provided 60 minute daily session.

General status of patients will be undertaken for the following outcomes at the baseline and 10 days after surgery (at discharge).

The primary outcome will be the visual analogue scale (VAS); the secondary outcomes will be: the disability knee assessed by the Western Ontario and McMaster Universities (WOMAC), the health related quality of life assessed by the EuroQol (EQ-5D), the global perceived effect assessed by the GPE score, the functional Independent measure assessed by the FIM questionnaire, the drugs assumption, the isometric strength of quadriceps and hamstrings assessed by dynamometer, the range of motion (R.O.M.) and proprioception assessed by VRRS.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral TKA for knee osteoarthritis
* informed consent

Exclusion Criteria:

* people with unstable serious disease (e.g., heart or lung disease)
* people with previous orthopedics pathologies on the same side (e.g., hip arthroprosthesis)
* pregnancy
* psychotropic drugs assumption

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Banfi, MD, Study Director — IRCCS Galeazzi Hospital
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

REFERENCES:
- [Derived] Gianola S, Stucovitz E, Castellini G, Mascali M, Vanni F, Tramacere I, Banfi G, Tornese D. Effects of early virtual reality-based rehabilitation in patients with total knee arthroplasty: A randomized controlled trial. Medicine (Baltimore). 2020 Feb;99(7):e19136. doi: 10.1097/MD.0000000000019136. PMID 32049833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Rehabilitation Department, IRCCS Orthopedic Institute Galeazzi, Milan, between September 2014 and November 2017.
Period: Overall Study
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Started | 44 | 41
Completed | 35 | 39
Not Completed | 9 | 2
Not completed — not comfortable with the intervention | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8.7) | 70.7 (8.5) | 69 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 24 | 13 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 41 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Right Total Knee Arthroplasty - no. (%) [Count of Participants; unit: Participants] | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Pain: Visual Analogue Scale (VAS)
Description: The VAS scale was measured in a range of 0-100 cm (0 no pain and 100 the worst pain)
Time Frame: baseline and 10 days (value at day 10 minus value at baseline)
Population: Available case analysis (drop-out <20%)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 35 | 39
units on a scale | -23.03 (21.06) | -28.97 (24.21)
Statistical Analysis 1: Comparison: VRRS Rehabilitation vs Traditional Rehabilitation; Does VRRS rehabilitation is superior to the traditional one?; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Net) = 5.94, 95% CI 2-sided [-4.62 to 16.51], Standard Deviation 5.30

2. Secondary Outcome: Knee Disability: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Questionnaire
Description: The WOMAC measures five items for pain (score range 0-500), two for stiffness (score range 0-200), and 17 for functional limitation (score range 0-1700) for a total score of 2400 (0= no disability, 2400= highest disability):
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties
Time Frame: baseline and 10 days (value at day 10 minus value at baseline)
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 35 | 39
units on a scale | 790.28 (234.36) | 767.6 (197.10)

3. Secondary Outcome: Knee Active Range of Motion
Description: assessed by Virtual Reality Rehabilitation System (degree of movement)
Time Frame: assesed and reported at 10 days
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 34 | 38
degree | 68.03 (13.56) | 69.75 (12.86)

4. Secondary Outcome: Health Related Quality of Life: Euro Quality of Life Five Dimensions Questionnaire (EQ-5D)
Description: The EQ-5D comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.The EQ-5D descriptive system is divided into five levels of perceived problems: LEVEL 1: indicating no problem; LEVEL 2:indicating some problems;LEVEL 3: indicating extreme problems. EQ-5D health states can be summarised using the 5-digit code (e.g., 11111, 12311).The answers given to ED-5D permit to find 243 5-digit codes defining the health states.The 5-digit code are linked to an unique index derived by applying a formula that attaches values (weights) to each of the levels in each dimension.Weights depend on the country (Italian Population-Based Values of EQ-5D HealthStates,Scalone 2013).The index has been calculated by deducting the appropriate weights from 1 which is the best health status as highest score (i.e. the corresponding 5-digit code is 11111) and -0.38 for the worst health status as minimum score (i.e., the corresponding 5-digit code is 33333).
Time Frame: assessed and reported at 10 days
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 35 | 39
units on a scale | 0.13 (0.11) | 0.15 (0.19)

5. Secondary Outcome: Global Perceived Effect (GPE)
Description: The GPE scale asks the patient to rate, on a numerical scale, how much their condition has improved or deteriorated since some predefined time point. The GPE was administered at the end of the physiotherapy treatment to measure the effect of the intervention on patients' health status perception. This Likert scale had five response options (5 = Very much improved; 4 = Much improved, 3 = No change, 2 = Much worse, 1 = Very much worse).
Time Frame: assessed and reported at 10 days
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 34 | 38
score on a scale | 4.58 (0.49) | 4.71 (0.45)

6. Secondary Outcome: The Functional Independence Measure (FIM) Scale
Description: The FIM scale assesses physical and cognitive disability focusing on the level of disability indicating the burden of caring for them. The total score is 126 (18=highest disability, 126=no disability).
Time Frame: baseline and 10 days (value at day 10 minus value at baseline)
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 35 | 39
units on a scale | 16.54 (9.23) | 20.10 (10.59)

7. Secondary Outcome: Proprioception
Description: assessed by Virtual Reality Rehabilitation System (percentage value of similarity between ideal and patient knee movement trajector)
Time Frame: assessed and reported at 10 day
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 33 | 38
mm | 73.46 (14.97) | 59.86 (19.85)

8. Secondary Outcome: Isometric Strength of Quadriceps and Hamstrings
Description: Isometric strength of quadriceps and hamstrings is assessed by dynamometer (newton unit)
Time Frame: baseline and 10 days (value at day 10 minus value at baseline)
Population: Available case analysis
Measure: Mean (Standard Deviation); unit: newton
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 28 | 30
newton | 25.08 (32.29) | 25.50 (28.98)

9. Secondary Outcome: Drugs Assumption
Description: number of drugs assumpted for each group during rehabilitation recovery
Time Frame: value at day 10
Population: descriptive
Measure: Number; unit: number of drugs assumpted per group
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
Number analyzed (Participants) | 35 | 39
number of drugs assumpted per group | 50 | 53

ADVERSE EVENTS:
Time Frame: 10 days after surgery
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | VRRS Rehabilitation | Traditional Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/44 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02413996/Prot_SAP_000.pdf